CLINICAL TRIAL: NCT01804426
Title: Hair Cortisol Level as a Predictor of PTSD Development
Status: Withdrawn | Type: Observational
Why Stopped: Lack of funding.
Sponsor: Shalvata Mental Health Center (Other)
Responsible Party: Principal Investigator, Aviv Segev, Psychiatry Resident, Shalvata Mental Health Center
Other Study IDs: MMC-12-221
Record Dates: First submitted 2013-02-28; First posted 2013-03-05 (Estimated); Last update posted 2016-04-20 (Estimated); Status verified 2016-04

CONDITIONS: Post Traumatic Stress Disorder
Keywords: PTSD; Post Traumatic Stress Disorder; Cortisol; Alpha-Amylase; bio-Markers
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — * Blood
  * Saliva
  * Hair
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Trauma Exposed participants: 18-50 years old men and women who have been brought to the ER after being involved or witnessing a life threatening event (or an event which was perceived as such).

SUMMARY:
Post-traumatic stress disorder, PTSD, is one of the most prevalent psychiatric disorders.

As casualties of motor vehicle accidents, criminal acts or terrorism are arriving to the ER, it is almost impossible to conclude who will overcome his psychiatric trauma and will be able to return to his normal life course and who will be thrown out of his promising life trajectory.

Current attempts to identify those who are at the greatest risk are still unsatisfactory, which comprise a therapeutic dilemma, since the interventions used to ameliorate and prevent the occurrence of PTSD in a high-risk patient, might be counter-productive and even precipitate the emergence of PTSD in lower-risk patients.

Since PTSD is closely related to the "Fight, Flight or Freeze" reaction, it has much to do with the autonomic nervous system and the major stress hormone, cortisol. Despite many studies demonstrating the involvement of those factors in the development of PTSD, various attempts to profile the direction of the association between PTSD and cortisol abnormalities have yielded conflicting results.

The introduction of a novel method of assessing the excretion of cortisol using residues in the human hair shaft, has allowed an unprecedented evaluation of its activity over a prolonged period of time.

Using this novel method of cortisol assessment, the investigators aim to identify biomarkers that will be able to aid in the prediction of PTSD development ahead of symptoms emergence, and will enhance the understanding of the physiological mechanism involved and etiology of this disorder.

DETAILED DESCRIPTION:
Post-Traumatic Stress Disorder (PTSD) stems from an event that is perceived as a threat to the physical and psychological integrity of the individual. Despite evidence pointing at predisposing or protective factors, it is extremely difficult to predict who will develop PTSD after exposure to a traumatic event. However, it is of a paramount importance to predict such a clinical course, in order to intervene at an early stage and facilitate research that may lead to prevention of the disorder.

As certain features of PTSD closely resemble the response of the adrenergic system via the fight or flight mechanism, substantial effort was made to understand the role of the hypothalamus-pituitary-adrenal (HPA) axis and the autonomic nervous system (ANS) in the development and maintenance of this disorder.

Various studies demonstrated conflicting findings, both in the trend of the level of cortisol and in the timing of the endocrinological anomaly. Additional study assessed the effect of HPA axis suppression by dexamethasone on anxiety-related symptoms in healthy volunteers subjected to a stress test. Those participants whose HPA axis was inhibited, presented a significant increase in anxiety symptoms, compared to a control group.

Variability and lack of stability are the main disadvantages of current methods quantifying systemic cortisol levels via measurements in the plasma, urine and saliva. These shortcomings undermine the effort to understand the role of the HPA axis in PTSD. Variable timing of the tests, as well as the stress involved in psychiatric examination and phlebotomy, are also major confounders in such an effort. Recently, the introduction of a novel test of hair cortisol concentration (HCC) has enabled retrospective quantification of cortisol levels, and thus the HPA axis activity, over a prolonged period of time.

As hair grows, unbounded cortisol is incorporated into the hair shaft in a manner that correlates with the amount of unbounded plasma cortisol at that time period. Since scalp hair grows at a fairly constant rate of 1cm per month, especially in the posterior vertex area, analysis of 3cm would reflect the average level of unbounded cortisol throughout the previous 3 months. Several studies in animals and humans have established the test's stability over time, thus proving that the test reliably reflects major changes in the HPA axis. Studies evaluating this novel test in the field of mental health demonstrated variations of cortisol levels in a number of clinical populations: increased hair cortisol levels were demonstrated for a 6 month period in depressed patients compared to controls; communities exposed to the horrors of war in Uganda had elevated cortisol levels compared to Ugandan communities not living in war zones; among patients with generalized anxiety disorder (GAD), there were lower hair cortisol levels in comparison with a control population, despite similar cortisol saliva levels.

In addition to the advantage of a reliable measurement of unbound plasma cortisol levels over time, this novel test is also easy to perform, easy to store and causes minimal inconvenience to the patient with no actual risks.

The use of this novel method of testing for cortisol level over prolong periods of time enables us to study the course of the HPA axis in relation to stressors: the baseline status, the immediate aftermath and the continuous effects of the traumatic event on the axis. Such valuable information can aid in the ongoing debate, whether the baseline function of the HPA axis is a core predisposing factor or, in fact, a secondary causality of the traumatic event.

Achieving better understanding of the complex interplay between those biological mechanisms and the formation of PTSD might enable the targeting of high-risk population after traumatic exposure with pharmacological and psychological interventions.

Study Hypothesis Main Hypothesis

1. Hair cortisol level previous to the trauma will correlate with PTSD development.

   Secondary Hypothesis
2. Ratio between hair cortisol levels prior to trauma to saliva cortisol level following the traumatic event will correlate with PTSD development.
3. Saliva cortisol level immediately after trauma will correlate with PTSD development.
4. Hair cortisol level one month post trauma will correlate with PTSD development.
5. Ratio between saliva cortisol levels to saliva alpha-amylase level (both taken at ER immediately after trauma) will correlate with PTSD development.
6. Patients with a difference between hair cortisol levels 3 months prior to the traumatic event and levels during the 3 months following it, are more prone to developing PTSD.

Study Methods Prospective observational study, performed at Meir Medical Center, Kfar Saba, Israel and Shalvata Mental Health Center, Hod Hasharon, Israel.

50 men and women arriving at Meir medical center Emergency department, as a result of a traumatic civil event, will be recruited.

Participants will fill out demographic and medical history questionnaires, and a structured psychiatric interview (M.I.N.I) will be performed to exclude any active psychiatric disorder. If none of the exclusion criteria met, several procedures will be performed:

1. Sampling hair from the posterior vortex.
2. Sampling blood cortisol and saliva cortisol and alpha-amylase.
3. Documenting pulse at the time of admission to the ER and 6 hours following the event.
4. Filling a number of questionnaires: SLE (stressful life events); BDI (Beck Depression Scale); MADRSS (Montgomery-Asberg Depression Rating Scale); STAI (State & Trait Anxiety Inventory); VAS-A, VAS-D; PDEQ (Peritraumatic Dissociation Experience Questionnaire); SASRQ (Stanford Acute Stress Reaction Questionnaire).

Psychiatric follow-up will be performed at 4 time points, in relation to the traumatic event: After 1 month, 3 months, 6 months and 12 months. During each assessment, the following procedures will be performed:

1. Sampling hair from the posterior vortex.
2. Filling out a number of questionnaires: BDI, MADRSS, STAI, VAS-A, VAS-D, CAPS (Clinician-Administered PTSD Scale), PSS (PTSD Symptoms Scale).

Relevance of potential study findings The proposed study will provide novel information on the role of the HPA axis in the development of PTSD. By answering this old, unresolved question the investigators will achieve an understanding of the neurobiological mechanism and may be able to predict the development of the disorder at an early, sub-clinical stage. The results of the study will also contribute to the understanding and rationale of the possibility of steroid treatment following an acute traumatic event.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-50
* Experienced a traumatic event fitting criterion A1 (stressor), A2 (Reaction) and at least 1 out of the B criterion in the ASD criteria in the DSM-IV-TR
* Brought to the ER within hours of the traumatic event.
* Signed an informed consent

Exclusion Criteria:

* Known psychiatric disorder or current psychiatric medication
* Complex injury or need for a complex medical treatment, such as operation, Packed RBC or admission extending 36 hours.
* Disorientation, confusion, head injury including intra-cranial bleeding, LOC or a major neurological deficit.
* Known disorder of the HPA axis or use of steroidal medications within the previous 3 years.
* known neurological disease or previous brain surgery.
* Major medical conditions or using medication known to influence the HPA or ANS Axis.
* Baldness or hair shorter than 1cm.
* Using color dyes.
* Pregnancy.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 50 men and women arriving at Meir medical center Emergency department, as a result of a traumatic civil event.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2013-03; Primary Completion 2015-07 (Estimated); Study Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in PTSD Symptoms | 3, 6, and 12 month post recruitment
  Change and development of PTSD symptoms from baseline using validated constructed psychiatric interview (CAPS) and self-administered questionnaire (PSS)

SECONDARY OUTCOMES:
ASD Development | 1 month
  Assessing development of Acute Stress Disorder, using the Stanford Acute Stress Reaction Questionnaire.
Change from Baseline in Hair Cortisol Levels | 1, 3, 6 and 12 months post recruitment
  Change in Hair Cortisol Levels from baseline at each of the assessment points (1, 3, 6 and 12 months).

CONTACTS AND LOCATIONS:
Overall Officials: Michael Lishner, MD, Prof, Principal Investigator — Meir Medical Center
Locations (1):
- Meir Medical Center, Kfar Saba, Israel